CLINICAL TRIAL: NCT02354274
Title: Novel Approach to Radiotherapy in Locally Advanced Lung Cancer - Heterogeneous FDG-guided Dose Escalation With Concomitant Navelbine®
Brief Title: Novel Approach to Radiotherapy in Locally Advanced Lung Cancer Concomitant Navelbine®
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Olfred Hansen (Other)
Collaborators: Odense University Hospital (Other); Aarhus University Hospital (Other); Rigshospitalet, Denmark (Other); Vejle Hospital (Other); Naestved Hospital (Other); Aalborg University Hospital (Other); Herlev Hospital (Other)
Responsible Party: Sponsor-Investigator, Olfred Hansen, MD, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NARLAL 2
Record Dates: First submitted 2015-01-19; First posted 2015-02-03 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: NSCLC

STUDY DESIGN:
Masking Description: Two independent radiation plans are made before randomization to ensure best available plans for both arms and trial.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard: Homogeneous dose plan (Active Comparator): Treatment will be given over 33 treatments. The dose is 66 Gy.
  Interventions: Radiation: Standard: Homogeneous dose plan
- Escalation: Inhomogeneous dose plan (Experimental): Radiation dose is increased to tumor and lymph nodes based on an inhomogeneous dose distribution determined by the most active ( FDG-PET criteria ) area of the node compared to a standard uniform dose distribution.
  Treatment will be given over 33 treatments. The dose is as high as possible taking the tolerance of the normal tissue into consideration
  Interventions: Radiation: Escalated: Inhomogeneous dose plan

INTERVENTIONS:
Radiation: Escalated: Inhomogeneous dose plan
  Arms: Escalation: Inhomogeneous dose plan
Radiation: Standard: Homogeneous dose plan
  Arms: Standard: Homogeneous dose plan

SUMMARY:
To investigate the effect of escalation of radiation dose to tumor and lymph nodes based on an inhomogeneous dose distribution controlled by FDG-PET positive areas compared to a standard homogeneous dose spread

DETAILED DESCRIPTION:
To investigate the effect of escalation of radiation dose to tumor and lymph nodes based on an inhomogeneous dose distribution controlled by FDG-PET-positive areas compared to a standard homogeneous dose spread.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically proven locally advanced NSCLC stage IIB to IIIB
* Performance status 0-1
* Able to comply with treatment and follow study and follow-up procedures
* Women must have negative pregnancy test
* Signed, informed consent
* Plan for radiotherapy with conventional 66 Gy/ 33 F, which meets all dosing limits two normal tissue must be available

Exclusion Criteria:

* Any unstable systemic disorder (including infection , unstable angina, congestive heart failure , severe liver , kidney or metabolic disease)
* Need for nasal oxygen
* Former thoracic radiotherapy, unless there is no significant overlap with previous fields
* Any other active malignant disease
* Unable to take oral medications or needing intravenous nutrition
* Ulcer
* Nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Locoregional control (Tumor recurrency is assessed by scheduled CT (of the thorax and upper abdomen) | 5-7 years
  Tumor recurrency is assessed by scheduled CT (of the thorax and upper abdomen ) every 3 months combined with PET/CT every 9 months or if occurrence is clinically suspected. Suspicion of tumor relapse local, regional or distant should be verified by biopsy. Date of detected recurrence is the date of the imaging modality suspecting relapse. The patient will be censured at death without local relapse.

SECONDARY OUTCOMES:
Toxicity (graded after CTCAE 4.0 assessed by physician) | 10 years
  Acute and late toxicity graded after CTCAE 4.0 assessed by physician at scheduled follow-up visits
Survival | 15 years
  Time from randomization to exact date of death of any cause.
Progression free survival | 15 years
  Time from randomization to date of progression, death, or occurence of metastatic disease

CONTACTS AND LOCATIONS:
Locations (7):
- Denmark (7):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Herlev University Hospital, Herlev
  - Department of Oncology, Naestved Hospital, Næstved
  - Department of Oncology, Odense University Hospital, Odense
  - Department of Oncology, Vejle Hospital, Vejle

REFERENCES:
- [Derived] Schytte T, Knap MM, Kristiansen C, Appelt AL, Khalil A, Peucelle C, Lutz CM, Moller DS, Sande EPS, Sundby F, Persson G, Schmidt H, Land LH, Rogg L, Pohl M, Lund MD, Nielsen M, Levin N, Hansen O, Thing RS, Borissova S, Halvorsen T, Nielsen TB, Hansen TS, Haakensen VD, Ottosson W, Brink C, Hoffmann L. Toxicity Within 6 Months of Heterogeneous Fluorodeoxyglucose-Guided Radiotherapy Dose Escalation for Locally Advanced Non-Small Cell Lung Cancer in the Scandinavian Randomized Phase III NARLAL2 Trial. J Clin Oncol. 2025 Jun 10;43(17):1972-1983. doi: 10.1200/JCO-24-01386. Epub 2025 Apr 18. PMID 40249893